CLINICAL TRIAL: NCT01578577
Title: EHR-based Health Literacy Strategy to Promote Medication Therapy Management
Brief Title: Northwestern University and Access Community Health Network Medication Education Study
Acronym: NAMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Medication Therapy Management; 1R01NR012745 (NIH)
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Hypertension
Keywords: Medication Therapy Management; Hypertension; Health Literacy; Medication Reconciliation; Medication Adherence
MeSH Terms: conditions — Hypertension; Medication Adherence | interventions — Faculty, Nursing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (No Intervention): This arm will serve as a control group and will not receive any intervention.
- EHMI (Experimental): Electronic Health Record-based Health Literacy Medication Therapy Management Intervention (EHMI)arm consists of multiple components, all leveraged by the Epic EHR platform (Verona, WI). The EHMI intervention 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides additional print tools to help patients more effectively engage their providers, consolidate their regimen, and generally promote safe use and adherence.
  Interventions: Behavioral: EHMI
- Nurse Educator + EHMI (Experimental)
  Interventions: Behavioral: Nurse Educator + EHMI

INTERVENTIONS:
Behavioral: EHMI — The EHMI intervention consists of multiple components, all leveraged by the Epic EHR platform (Verona, WI). The EHMI intervention 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides additional print tools to help patients more effectively engage their providers, consolidate their regimen, and generally promote safe use and adherence.
  Arms: EHMI
Behavioral: Nurse Educator + EHMI — This intervention is a combination of the use of a nurse educator and the EHMI tools described in the EHMI intervention arm. A nurse educator perform the following: 1) perform medication and medical record review 2)assess adherence and medication problems 3) provide counseling to promote safe and effective medication use 4) follow-up with patients after their visit to confirm they have filled all prescriptions, and can accurately teach back their medicine regimen, 5) communicate with prescribing physician when problems are identified.
  Arms: Nurse Educator + EHMI

SUMMARY:
Many patients have difficulty performing routine medication management tasks. Individuals with limited literacy are at high risk for these problems. The overall study objective is to rigorously evaluate two primary care-based medication therapy management strategies that leverage an electronic health record (EHR) to promote patient understanding, medication reconciliation, medication adherence and disease control among hypertensive patients at safety net clinics.

DETAILED DESCRIPTION:
Medication therapy management (MTM) has been described as a set of procedures that include: medication review, assembly of a personal medication record, development of action plans, intervention when necessary, and follow-up. However, evidence showing the effectiveness of general MTM interventions is scant. MTM has often been performed separately from patients' usual sources of care (i.e., at pharmacies). This could limit its effectiveness since medication-related concerns would be discussed by clinicians who are not aware of the regimen intended by patients' prescribers. Cost is another barrier to widespread use of MTM.

Health information technology in primary care could be leveraged to assist with MTM tasks. The investigators have field tested low literacy MTM tools embedded within an EHR to 1) activate patients to review medications, 2) automate the provision of plain language, medication information, and 3) provide print tools to help patients engage providers, and consolidate their regime. These tools were developed with patient, physician, and pharmacist feedback.

For this study, the investigators combine tools to address the range of MTM tasks. In aggregate, the study refers to this as an Electronic health record-based Health literacy Medication therapy management Intervention, or 'EHMI'. The investigators will evaluate the effects of this approach among patients with uncontrolled hypertension treated in federally qualified health centers (FQHCs). This may be a relatively low-cost strategy ideal for safety net practices that use EHRs and whose patients may be at greater risk for limited literacy. It is also possible that the EHMI strategy may not result in a significant change. Therefore, the investigators will also evaluate using a nurse educator to help patients utilize EHMI tools, provide brief counseling, and track progress.

This three-arm, clinic-randomized, controlled trial conducted within a network of FQHCs will evaluate the EHMI and EHMI + Nurse Educator interventions compared to usual care. Recruited patients will be followed for 12 months. The investigators will test the impact of these two strategies on blood pressure levels, with an anticipated power to detect a 4 mm Hg difference in systolic blood pressure as the primary outcome. The investigators will also assess the impact on diastolic blood pressure, as well as HbA1c and LDL cholesterol control in the subgroup with diabetes. The investigators will determine the interventions' effects on: 1) medication understanding, 2) discrepancies, and 3) adherence. The investigators will specifically examine intervention effects among groups with different literacy levels. The investigators will also assess the fidelity and cost of the interventions to guide future dissemination efforts.

ELIGIBILITY:
Inclusion Criteria:

* age is 18 years or older
* at least 3 medications are prescribed by their physician
* standardized mean blood pressure measurement ≥130 mm Hg systolic or ≥ 80 mm Hg diastolic if they are diabetic or mean blood pressure measurement ≥ 135 mm Hg systolic or ≥ 85 mm Hg diastolic if they are not
* a Mini-Cog Exam score of ≥ 3
* the patient is the person primarily responsible for administering their medication
* the patient does not intend to move or change their usual source of medical care during the next year.

Exclusion Criteria:

* the patient's usual source of medical care is not a participating ACCESS Community Health Center
* is non-English language speaking
* does not meet mean blood pressure criteria
* has a Mini-Cog Exam score of < 3
* is not the person primarily responsible for administering medication
* intends to move or change their usual source of medical care during the next year.
* Is not prescribed at least 3 medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 920 (Actual)
Dates: Start 2012-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Persell, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- ACCESS Community Health Network, Chicago, Illinois, United States

REFERENCES:
- [Derived] Persell SD, Karmali KN, Lazar D, Friesema EM, Lee JY, Rademaker A, Kaiser D, Eder M, French DD, Brown T, Wolf MS. Effect of Electronic Health Record-Based Medication Support and Nurse-Led Medication Therapy Management on Hypertension and Medication Self-management: A Randomized Clinical Trial. JAMA Intern Med. 2018 Aug 1;178(8):1069-1077. doi: 10.1001/jamainternmed.2018.2372. PMID 29987324
- [Derived] Persell SD, Eder M, Friesema E, Connor C, Rademaker A, French DD, King J, Wolf MS. EHR-based medication support and nurse-led medication therapy management: rationale and design for a three-arm clinic randomized trial. J Am Heart Assoc. 2013 Oct 24;2(5):e000311. doi: 10.1161/JAHA.113.000311. PMID 24157649

RESULTS

PARTICIPANT FLOW:
Groups:
- EHMI: Electronic Health Record-based Health Literacy Medication Therapy Management Intervention (EHMI)arm consists of multiple components. The EHMI intervention 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides additional print tools to help patients more effectively engage their providers, consolidate their regimen, and generally promote safe use and adherence.
  EHMI: The EHMI intervention consists of multiple components, all leveraged by the Epic EHR platform (Verona, WI). The EHMI intervention 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides
Period: Overall Study
Arm/Group | Standard Care | EHMI | Nurse Educator + EHMI
Started | 305 | 302 | 313
Completed | 254 | 262 | 278
Not Completed | 51 | 40 | 35

BASELINE CHARACTERISTICS:
Groups:
- EHMI: Electronic Health Record-based Health Literacy Medication Therapy Management Intervention (EHMI)arm consists of multiple components. The EHMI 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides additional print tools to help patients more effectively engage their providers, consolidate their regimen, and generally promote safe use and adherence.
- Total: Total of all reporting groups
Arm/Group | Standard Care | EHMI | Nurse Educator + EHMI | Total
Number analyzed (Participants) | 254 | 262 | 278 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (9.5) | 53.6 (9.7) | 51.6 (9.5) | 52.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 175 | 187 | 545
  Male | 71 | 87 | 91 | 249
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 23 | 37
  Not Hispanic or Latino | 237 | 250 | 233 | 720
  Unknown or Not Reported | 7 | 8 | 22 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 234 | 243 | 215 | 692
  White | 13 | 11 | 41 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 22 | 37

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: The primary outcome is the systolic blood pressure measured approximately one year after the baseline interview is conducted.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Standard Care | EHMI | Nurse Educator + EHMI
Number analyzed (Participants) | 254 | 262 | 278
mm Hg | 134.5 (20.4) | 141.7 (22.1) | 134.6 (19.9)

2. Secondary Outcome: Effectiveness of the Electronic Health Record-based Health Literacy Medication Therapy Management Strategy (EHMI), With and Without a Nurse Educator, Compared to Standard Care.
Description: This will be assessed by measuring patient medication understanding, medication reconciliation, adherence, and health outcomes (diastolic blood pressure, and among the diabetic subgroup Hemoglobin A1c <8.0 and LDL Cholesterol <100).
  Reported here: HbA1c <8 at 12 months. Full secondary outcomes have been published. Persell SD, Karmali KN, MD, Lazar D, Friesema EM, Lee JY, Rademaker A, Kaiser D, Eder M, French DD, Brown T, Wolf MS. Effect of electronic health record-based medication support and nurse-led medication therapy management on hypertension and medication self-management: a randomized clinical trial. JAMA Intern Med. 2018;178:1069-1077.
Time Frame: Baseline, 3 months, 6 months, 12 months
Measure: Count of Participants; unit: Participants
Groups:
- EHMI: EHMI: The EHMI intervention consists of multiple components. The EHMI intervention 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides
Arm/Group | Standard Care | EHMI | Nurse Educator + EHMI
Number analyzed (Participants) | 130 | 111 | 107
Participants | 61 | 48 | 64

3. Secondary Outcome: Effects of These Strategies by Patients' Literacy Skills
Description: We will measure how the effects of the interventions vary based on the participants' literacy levels.
  SBP at 12 months reported below.
Time Frame: Baseline, 3 months, 6 months,12 months
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Standard Care Likely Limited Health Literacy: This arm will serve as a control group and will not receive any intervention.
- EHMI Likely Limited Health Literacy: EHMI: The EHMI intervention consists of multiple components. The EHMI intervention 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides
- Nurse Educator + EHMI Likely Limted Health Literacy: Nurse Educator + EHMI: This intervention is a combination of the use of a nurse educator and the EHMI tools described in the EHMI intervention arm. A nurse educator perform the following: 1) perform medication and medical record review 2)assess adherence and medication problems 3) provide counseling to promote safe and effective medication use 4) follow-up with patients after their visit to confirm they have filled all prescriptions, and can accurately teach back their medicine regimen, 5) communicate with prescribing physician when problems are identified.
- Standard Care Possibly Limited Health Literacy: Standard Care Possibly Limited Health Literacy
- EHMI Possibly Limited Health Literacy: EHMI Possibly Limited Health Literacy
- Standard Care Likely Adequate Health Literacy: Standard Care Likely Adequate Health Literacy
- EHMI Likely Adequate Health Literacy: EHMI Likely Adequate Health Literacy
- Nurse Educator + EHMI Likely Adequate Health Literacy: Nurse Educator + EHMI Likely Adequate Health Literacy
Arm/Group | Standard Care Likely Limited Health Literacy | EHMI Likely Limited Health Literacy | Nurse Educator + EHMI Likely Limted Health Literacy | Standard Care Possibly Limited Health Literacy | EHMI Possibly Limited Health Literacy | Nurse Educator + EHMI Possibly Limited Health Literacy | Standard Care Likely Adequate Health Literacy | EHMI Likely Adequate Health Literacy | Nurse Educator + EHMI Likely Adequate Health Literacy
Number analyzed (Participants) | 145 | 126 | 104 | 75 | 90 | 98 | 34 | 46 | 76
mm Hg | 135.5 (20.7) | 141.7 (20) | 133.8 (18.8) | 138.4 (22.4) | 138.4 (22.4) | 132.2 (19.4) | 135.5 (20.1) | 148.1 (25.7) | 138.9 (21.5)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Note, this study did not include a systematic collection of adverse events. No adverse events related to the study procedures were reported.
Groups:
- EHMI: EHMI: The EHMI intervention consists of multiple components, all leveraged by the Epic EHR platform (Verona, WI). The EHMI intervention 1) activates patients to review their medication list and identify any adherence-related concerns, 2) automates a process for providing plain language, patient-centered print medication information for new and refilled prescriptions, and 3) provides
Arm/Group | Standard Care | EHMI | Nurse Educator + EHMI
Serious Adverse Events (participants affected / at risk) | 0/305 | 0/302 | 0/313
Other Adverse Events (participants affected / at risk) | 0/305 | 0/302 | 0/313

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No